CLINICAL TRIAL: NCT06329167
Title: Clinical Trial of Daphnetin Capsules for Lower Limb Lymphoedema Following Gynaecological Surgery
Brief Title: Daphnetin Capsules for Lower Limb Lymphoedema Following Gynaecological Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Songling Zhang, vice president, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-HS-012
Record Dates: First submitted 2024-03-11; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Lower Extremity Lymphedema
Keywords: Lower Extremity Lymphedema; gynaecological malignancy surgery; daphnetin; Aescuven
MeSH Terms: interventions — daphnetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daphnetin treatment group (Experimental): Daphnetin capsule 150mg tid (3 capsules/time, 3 times daily) and gradient compression stockings.
  Interventions: Drug: Daphnetin
- Aescuven Forte group (Active Comparator): Aescuven Forte oral tablet 150mg (2 capsules/time, 2 times daily) and gradient compression stockings.
  Interventions: Drug: Aescuven

INTERVENTIONS:
Drug: Daphnetin — 150mg tid (3 capsules/time, 3 times daily) and gradient compression stockings.
  Other Names: gradient compression stocking
  Arms: Daphnetin treatment group
Drug: Aescuven — 150mg (2 capsules/time, 2 times daily) and gradient compression stockings.
  Other Names: gradient compression stocking
  Arms: Aescuven Forte group

SUMMARY:
This clinical trial is designed to learn more about treating patients with lower limb lymphoedema following gynaecological surgery. The main question to be answered is To evaluate the efficacy of Daphnetin capsule in the treatment of patients with lower limb lymphedema following gynaecological malignancy surgery. Participants will take Daphnetin capsule 150mg tid (3 capsules/time, 3 times daily) orally at the same time as gradient compression stocking treatment. Researchers will compare 150mg Forte tablets (2 capsules/time, 2 times daily) and gradient compression stockings to see if Daphnetin capsule can be used to treat patients with lower extremity lymphedema following gynaecological malignancy surgery.

DETAILED DESCRIPTION:
This study was a randomised, controlled, open-label, single-centre clinical trial. The objective of this study was to determine the efficacy and safety of Daphnetic capsules compared to Aesculete tablets in the treatment of patients with lower extremity lymphedema following gynaecological cancer surgery. A total of 100 patients with postoperative lower extremity lymphedema (stage I-II) following gynaecological cancer surgery were enrolled in this randomised controlled trial. Patients were randomised 1:1 to the experimental or control group.

Subjects who met the inclusion and exclusion criteria were randomly allocated to the Daphnetin group (study group) or the Aesculeum aesculeum group (control group) in a 1:1 ratio after signing the informed consent form. Both groups were treated for 21 days as a cycle, and efficacy and safety indices were evaluated after the first course of treatment.

Group A: Daphnetin capsule 150mg tid (3 capsules/time, 3 times daily) and gradient compression stockings.

Group B: Aescuven Forte oral tablet 150mg (2 capsules/time, 2 times daily) and gradient compression stockings.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years (including cut-off) with lower limb lymphoedema (stage I-II) following gynaecological surgery for a malignant tumour without temporary surgical treatment.
* There was no preoperative lymphedema
* Voluntarily sign consent form
* The performance status score had to be 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG).
* Investigator-assessed expected survival ≥12 weeks
* Not receiving any other treatment for lower limb lymphoedema
* Have adequate organ and bone marrow reserve function
* Be able to understand the requirements of the trial and be willing and able to follow the trial and follow-up procedures

Exclusion Criteria:

* A history of severe trauma to the lower limbs;
* Diseases that can cause lower limb oedema such as primary lymphatic disease, venous thrombosis, cardiogenic, nephrogenic, hypoproteinemia and other systemic diseases that can cause lower limb oedema.
* Colour Doppler ultrasonography of the lower limbs suggesting lower limb vascular disease;
* Patients with a history of allogeneic cell or solid organ transplantation;
* primary central nervous system tumour or symptomatic central nervous system metastasis, meningeal metastasis, or history of epilepsy. Patients with clinically controlled CNS metastases that were asymptomatic or symptomatic but stable in the opinion of the investigators were eligible if the following conditions were met: a. Clinical symptoms were stable for more than 4 weeks prior to the first dose; b. No evidence of CNS disease progression on contrast-enhanced MRI of the head within 4 weeks prior to the first dose; c. Prednisone ≤10 mg/day or equivalent hormone dose was discontinued at least 2 weeks prior to the first dose of antiepileptic drugs.;
* other active malignancies within 5 years prior to the first dose. Except for locally cured tumours (such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder carcinoma, or carcinoma in situ of the breast);
* Any of the following cardiovascular diseases occurring within 6 months prior to the first dose of the drug: symptomatic heart failure of New York Heart Association (NYHA) class 2 or higher, left ventricular ejection fraction (LVEF) less than 50%, unstable arrhythmia, or unstable angina, Myocardial infarction requiring treatment, pulmonary embolism, or uncontrolled hypertension, defined in this protocol as systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg after treatment and clinically significant as assessed by the investigator);
* The presence of any other medical condition, physical examination, or laboratory test results that, in the opinion of the investigator, are unsuitable for use of the study drug;
* combined with long-term oral vitamin K disease
* Subjects with untreated or treated tuberculosis, including but not limited to tuberculosis; patients who received standard anti-tuberculosis treatment and were confirmed cured by the investigators were eligible.
* Severe infection had occurred within 4 weeks or active infection had occurred within 2 weeks prior to the first medication;
* Patients with the following diseases: human immunodeficiency virus (HIV) infection; active hepatitis B virus infection [hepatitis B surface antigen (HBsAg) positive and hepatitis B virus DNA (HBV DNA) >200 IU/mL or 103 copies/mL]; hepatitis C virus infection (HCV antibody and viral RNA (HCV RNA) test results were positive); patients with Treponema pallidum antibody positive and RPR positive;
* Known hypersensitivity or delayed allergic reaction to any component of the study drug;
* Known history of mental disorders, drug abuse, alcoholism, or substance abuse that may affect the test results;
* the patient's lack of compliance to participate in the clinical trial or the presence of any other factor that the investigator deems inappropriate for participation in the trial.
* patients with tumour recurrence or metastasis during follow-up.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female after gynaecological malignancy surgery
Enrollment: 100 (Estimated)
Dates: Start 2024-03-25 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
The difference in the circumference of the lower limbs | day 14, day 21, day 28
  The patient was in the supine position with both lower limbs relaxed. The clinician measured the limb circumference at the dorsum of the foot, the lateral malleolus, the upper edge of the patella and 10 cm above and below with a tape measure and calculated the difference in limb circumference between the two lower limbs.
Gynaecological Cancer Lymphedema Questionnaire | day 14, day 21, day 28
  The GCLQ has good reliability and validity and is easy to administer. It is widely used in the diagnosis and assessment of lower extremity lymphoedema. The questionnaire consisted of 20 questions scored on 7 dimensions: heaviness, oedema (global), swelling (local), numbness, infection, pain and limb function. The answer 'yes' to each question was worth 1 point and the answer 'no' was worth 0 point. A total score of ≥4 points was considered to be lower limb lymphedema (see Appendix II).
Fibrinogen content | day 14, day 21, day 28
  2ml of peripheral venous blood was collected from patients and stored in EDTA anticoagulant test tubes. FIB was detected by automatic haemagglutination analyser (STAGO MAXR) in the laboratory department of our hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- the 1st hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No